CLINICAL TRIAL: NCT05277129
Title: The Immune Response to Stroke
Status: Recruiting | Type: Observational
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Andreas Lossius, Associate Professor, University of Oslo
Other Study IDs: 2019/1252
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Stroke, Acute; Dementia
MeSH Terms: conditions — Stroke; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients
  Interventions: Other: Analysis of post-stroke immune responses

INTERVENTIONS:
Other: Analysis of post-stroke immune responses — Analysis of immune responses in peripheral blood

SUMMARY:
Some patients develop cognitive decline after a stroke, but we don't always understand the mechanisms. It has been proposed that a proportion of the patients develop an autoimmune immune response, and that this could potentially explain the cognitive decline in some of the patients. The current study aims to investigate this hypothesis in a subgroup of patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

* Stroke < 72 h
* Age > 18 years

Exclusion Criteria:

* Brain hemorrhage verified by CT or MRI scan
* Previous or present immunological disease or other serious comorbidity
* Ongoing immune respons after infection or vaccination < 1 month
* Cognitive without ability to understand and/or give an informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from acute cerebral infarction
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-06-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-06-06 (Estimated)

PRIMARY OUTCOMES:
The B cell and T cell response in peripheral blood | 1 day (subject inclusion)

CONTACTS AND LOCATIONS:
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No